CLINICAL TRIAL: NCT00364078
Title: Transitoriness in Cancer Patients: a Cross-Sectional Study of Uncertainty, Locus of Control, Quality of Life and Existentials Views on Finality of Life in Cancer Patients
Brief Title: Transitoriness in Cancer Patients, Psychosocial Issues in Cancer Care
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Swiss Cancer League (Other); Johns Hopkins University (Other)
Responsible Party: Maya Shaha, PhD, Johns Hopkins University School of Nursing
Other Study IDs: J0601; BIL OCS 01532-03-2004; Dorothy Evans Lyne Fund
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Lung Cancer; Gastrointestinal Cancers
Keywords: Cross-sectional correlational study; Uncertainty; Locus of Control; Quality of life; Transitoriness; Cancer care
MeSH Terms: conditions — Lung Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Transitoriness can be defined as confrontation with life's finitude. Cancer patients are perceived to experience this confrontation due to their diagnosis. It is perceived to impact cancer patients' ways of coping with the disease situation. In this study, cancer patients' levels of uncertainty, transitoriness and their perceived locus of control are assessed. It is aimed at exploring the association of uncertainty, locus of control, transitoriness and quality of life. If a stronger correlation of one or the other issue with quality of life can be discovered, it will inform the development of an adequate evidence-based nursing intervention to better support patients' coping with the disease.

DETAILED DESCRIPTION:
Cancer is the second leading cause of death among individuals in the United States of America (Ries et al., 2000). Gastro-intestinal (GI) cancers account for approximately 253,500 new cases each year in both men and women. Most of the patients with GI cancer have a poor outcome (American Cancer Society., 2005; Ilson, 2001), accounting for approximately 16% of cancer related death in women and 25% of cancer related death in men (American Cancer Society, 2005). Of all cancers, lung cancer is the leading cause for death among men and women (American Cancer Society., 2005).

GI cancer constitutes a disease with intensive medical research focused on the improvement of prevention, early detection and treatment. How patients with GI cancer deal with the diagnosis remains understudied to date. Lung cancer research has focused particularly on smoking and its impact on lung cancer epidemiology. Lung cancer patients' coping strategies have been studied. Issues related to the meaning of life, health and self-care, physical functioning, coping and support have been highlighted as being important in lung cancer patients' dealing with their disease situation (Maliski, Sarna, Evangelista, & Padilla, 2003; Sharf, Stelljes, & Gordon, 2005). Similarly, patients' dealing with a diagnosis of breast cancer has been investigated (Andritsch et al., 2004; Badger, Braden, Mishel, & Longman, 2004; Northouse, Templin, Mood, & Oberst, 1998). Constructs such as uncertainty and locus control are highly important in coping with the disease situation. Uncertainty has been linked with quality of life (Sammarco, 2001;2003). Evidence also exists that transitoriness, which is the confrontation with the finitude of human life, plays an important role in how individuals cope (Cohen et al., 2004; Shaha & Cox, 2003). The interrelationship between and among transitoriness, uncertainty and locus of control has yet to be delineated. There is also a need to explore transitoriness more fully as it has mainly been subsumed in concepts such as 'finding meaning in illness' or 'anxiety' (Houldin, 2003). Transitoriness has been linked with patient outcomes such as quality of life (Houldin, 2003). It is necessary to explore the concept of transitoriness to establish its links with uncertainty and locus of control. It is equally important to explore the association of these three concepts together with patients' psycho-social well-being and quality of life. By exploring these associations, the individual's way of coping with the cancer diagnosis will be better understood and lead to the development of nursing interventions to support persons with cancer, especially those with lung and GI cancer.

It will then be possible a) to explore the concept of transitoriness by describing its interrelationship with uncertainty and locus of control, and b) to investigate the association among transitoriness, uncertainty, locus of control, psycho-social well-being and quality of life. The following research questions will be addressed in the study:

1. Is cancer patients' confrontation with life's finitude related to uncertainty and locus of control?
2. Are cancer patients' confrontation with life's finitude, uncertainty and locus of control associated with psychosocial well-being and quality of life?
3. Are there differences in these associations between patients with different forms of cancer?

ELIGIBILITY:
Inclusion Criteria:

* Lung and gastrointestinal cancer diagnoses at various stages
* Inpatient or outpatient of Johns Hopkins Hospital, Sidney Kimmel Cancer Center, Bayview Medical Center or Greensprings Station
* Ability to read and understand English
* 18 years or older
* Patients have been informed of the serious/terminal nature of their cancer diagnosis
* Physically and mentally fit
* Diverse ethnic background

Exclusion Criteria:

* Observable evidence of confusion (researcher will consult with psychiatric liaison nurse if the patient is not oriented to time,place and person).
* Patients who experience pain or other discomforting symptoms
* Receiving hospice care

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Johns Hopkins University Medical Institutions
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Belcher, PhD, Principal Investigator — Johns Hopkins School of Nursing
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

REFERENCES:
- [Background] Shaha M, Cox CL. The omnipresence of cancer. Eur J Oncol Nurs. 2003 Sep;7(3):191-6. doi: 10.1016/s1462-3889(03)00026-7. PMID 12932481
- [Background] Shaha M. [Life with intestinal cancer. A phenomenologic-empirical study]. Pflege. 2003 Dec;16(6):323-30. doi: 10.1024/1012-5302.16.6.323. German. PMID 14964130
- [Background] Shaha M, Cox C, Porrett T, Hall A.The omnipresence of cancer and its practice implications for colorectal cancer. Cancer Nursing Practice, 5(4): 35 - 39, 2006
- [Background] Shaha M, Cox CL, Talman K, Kelly D. Uncertainty in breast, prostate, and colorectal cancer: implications for supportive care. J Nurs Scholarsh. 2008;40(1):60-7. doi: 10.1111/j.1547-5069.2007.00207.x. PMID 18302593